CLINICAL TRIAL: NCT04518189
Title: Transdermal Lidocaine for Pain Control During Hysterosalpingography: A Randomized Controlled Trial
Brief Title: Transdermal Lidocaine for Pain Control During Hysterosalpingography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, A Professor, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu/295/3/19
Record Dates: First submitted 2020-08-15; First posted 2020-08-19 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Intervention Model Description: double blind randomized trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lidocaine patch (Experimental): 5% lidocaine patch applied at 3 hours before the procedure
  Interventions: Drug: lidocaine patch
- Sham patch (Placebo Comparator): Sham patch containing no study medication applied 3 hours before the procedure
  Interventions: Drug: Sham patch

INTERVENTIONS:
Drug: lidocaine patch — lidocaine patch applied 3 hours before the procedure
  Other Names: Experimental
  Arms: lidocaine patch
Drug: Sham patch — Sham patch applied 3 hours before the procedure
  Other Names: Placebo Comparator
  Arms: Sham patch

SUMMARY:
the study aims to investigate the effectiveness of Transdermal lidocaine patch for Pain Control During Hysterosalpingography

DETAILED DESCRIPTION:
hysterosalpingography can cause pain and discomfort in several ways: Use of the tenaculum to grasp the cervix and straighten the uterus for proper insertion; trans-cervical actions including measuring uterine depth, inserting the cannula; and injection of the dye

ELIGIBILITY:
Inclusion Criteria:

* any patient came for Hysterosalpingography

Exclusion Criteria:

* any patient has contraindication to Hysterosalpingography

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — any patient came for Hysterosalpingography
Enrollment: 120 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Mean pain score during the procedure | 10 minutes
  Assessment of pain using visual analog scale 0-10, 0 = minimum and 10 = maximum scores

CONTACTS AND LOCATIONS:
Overall Officials: nahla w Shady, md, Study Chair — Aswan universirty
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No